CLINICAL TRIAL: NCT01207700
Title: A Randomized, Open Trial Comparing Post Discharge Interventions to Standard Care
Brief Title: Secondary Prevention of coRonary Events After Discharge From Hospital (SPREAD)
Acronym: SPREAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Collaborators: National Heart and Lung Institute (Other)
Responsible Party: Principal Investigator, Dr Alben Sigamani, Associate Professor, St. John's Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NO1-HV-98215/SJRI - DCT/SPREAD
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Acute Coronary Syndrome
Keywords: post discharge intervention; adherence; compliance; community health worker
MeSH Terms: conditions — Acute Coronary Syndrome; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHW based intervention post ACS (Experimental): CHW trained and supervised for intervening upon post ACS patients to improve adherence to evidence based care
  Interventions: Behavioral: CHW based intervention post ACS
- Standard Care (No Intervention): Patients will be followed upto 12 months without a community health worker intervention as per standard practices of the hospital

INTERVENTIONS:
Behavioral: CHW based intervention post ACS — CHW is trained and supervised to provide interventions that could improved adherence to post ACS care
  Arms: CHW based intervention post ACS

SUMMARY:
This is a randomized, open trial comparing post discharge interventions by community health workers (CHW) to standard care in acute coronary syndrome (ACS) patients.

This trial will be conducted in 10 hospitals in India/different parts(both secondary and tertiary care). A total of 800 patients will be recruited, with equal allocation to SPREAD interventions and control groups (usual care)

DETAILED DESCRIPTION:
Inclusion criteria:

Consenting patients being discharged after an acute coronary event such as unstable angina, acute myocardial infarction, or after coronary intervention (CABG surgery or PCI).

Exclusion criteria:

Patients with other terminal/ debilitating illness, (e.g., advanced cancer, disabling stroke) those not expected to survive for the study duration, those with dementia and psychiatric illness or patients unlikely to comply with study requirements, including regular follow up.

OUTCOME MEASURES:

1. Feasibility
2. Difference in adherence to specific medications for secondary prevention of CAD (Coronary Artery Diseases) compared to the control group, at one year.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients being discharged after an acute coronary event such as unstable angina, acute myocardial infarction, or after coronary intervention (CABG surgery or PCI).

Exclusion Criteria:

* Patients with other terminal/ debilitating illness, (e.g., advanced cancer, disabling stroke) those not expected to survive for the study duration, those with dementia and psychiatric illness or patients unlikely to comply with study requirements, including regular follow up

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To obtain estimates of rates of adherence to pharmacotherapy and lifestyle modification interventions and the incidence of major cardiovascular events | 12 months
  Evaluate the rates of adherence to pharmacotherapy and lifestyle modifications using the community health worker
To determine the feasibility of conducting a secondary prevention trial using CDCHWs on adherence to medications and lifestyle advice | 12 MONTHS
  A pilot study to look at feasibiility of using a trained community health worker to deliver health messages to patients who have had a coronary event

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rajeev Gupta, MD, PHD, Principal Investigator — Fortis Escorts Hospital, Jaipur
Locations (13):
- India (13):
  - Krishna Institute of Medical Science Ltd, Secunderabad, Aandhra Pradesh
  - Mahavir Hospital & Research Centre, Hyderabad, Andhra Pradesh
  - Nanjappa Hospital, Shimoga, Karnataka
  - Caritas Hospital, Kottayam, Kerala
  - Bhopal Memorial Hospital, Bhopal, Madhya Pradesh
  - Avanti Institute of Cardiology, Nagpur, Maharashtra
  - Poona Hospital, Pune, Maharashtra
  - Mahatma Gandhi Institute of Medical Science Sevagram, Wardha, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, New Delhi
  - Fortis Escorts Hospital, Jaipur, Rajasthan
  - Rajamuthiah Medical College & Hospital, Annāmalainagar, Tamil Nadu
  - PSG Hospital, Coimbatore, Tamil Nadu
  - Sahara Hospital, Lucknow, Uttar Pradesh

REFERENCES:
- [Derived] Xavier D, Gupta R, Kamath D, Sigamani A, Devereaux PJ, George N, Joshi R, Pogue J, Pais P, Yusuf S. Community health worker-based intervention for adherence to drugs and lifestyle change after acute coronary syndrome: a multicentre, open, randomised controlled trial. Lancet Diabetes Endocrinol. 2016 Mar;4(3):244-253. doi: 10.1016/S2213-8587(15)00480-5. Epub 2016 Feb 6. PMID 26857999